CLINICAL TRIAL: NCT02473315
Title: Assessment of Whole Body Cryotherapy in Treatment of Active Axial Spondylarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015- A00337-42
Record Dates: First submitted 2015-06-10; First posted 2015-06-16 (Estimated); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Spondylarthritis
MeSH Terms: conditions — Spondylarthritis | interventions — Cryotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- cryotherapy (Experimental)
  Interventions: Other: cryotherapy
- light cryotherapy (Placebo Comparator)
  Interventions: Other: cryotherapy

INTERVENTIONS:
Other: cryotherapy — The treatment arm :Whole body cryotherpy (WBC) (20 sessions of 3 minutes at a temperature of -110 degrees Celsius, on the basis of two sessions a day, spread over two weeks).
  The control arm : Whole body cryotherpy (WBC) (20 sessions of 1 minute at a temperature of -60 degrees Celsius, on the basis of two sessions a day, spread over two weeks).

SUMMARY:
Whole body cryotherpy (WBC) is a well-tolerated procedure that implies patients' exposition at a temperature of approximately -110 degrees.

A considerable increase in the popularity of WBC has occurred in rheumatologic patients, despite a lack of evidences of its efficiency.

Because of its interesting anti-inflammatory properties, the investigators think that WBC could be an alternative treatment to classical NSAIDs (Non Steroidal Anti Inflammatory Drugs) and corticosteroids, in patients suffering from axial spondyloarthritis.

This is a proof of concept study.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from axial spondyloarthritis diagnosed according to ASAS criteria, with sacroiliitis on X-rays or MRI, with active disease (BASDAI > 4/10) despite a stable treatment will be included.

Exclusion Criteria:

* contra indication to cooling,
* previous WBC treatment,
* no social security cover

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-09-18 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
Whole body cryotherpy (WBC) efficacy assesment | 15 days
  assess WBC efficacy on disease activity with Bath Ankylosing Spondylitis Activity Index improvement between baseline and week 2 in patients with active axial spondyloarthritis. a difference of 20 points on BASDAI scale is expected between the experimental arm and the placebo is expected

CONTACTS AND LOCATIONS:
Overall Officials: ANNA DELLYES, MD, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France